CLINICAL TRIAL: NCT06686615
Title: Effectiveness and Safety of Bempedoic Acid in Combination With Ezetimibe and Either Rosuvastatin or Atorvastatin in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia: an Observational Study
Brief Title: A Study of Bempedoic Acid in Combination With Ezetimibe and Either Rosuvastatin or Atorvastatin in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Acronym: TRICONOS
Status: Recruiting | Type: Observational
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DSE-BMP-01-24-EU
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Primary Hypercholesterolemiia; Mixed Dyslipidemia
Keywords: Primary hypercholesterolemia; Mixed dyslipidemia
MeSH Terms: interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe; Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triple therapy: Adult patients who have been diagnosed with primary hypercholesterolaemia (heterozygous familial and nonfamilial) or mixed dyslipidaemia treated with bempedoic acid in combination with ezetimibe and either rosuvastatin or atorvastatin (ie, triple therapy) and will be followed for up to 1 year after initiation of triple therapy.
  A direct comparison between rosuvastatin and atorvastatin is not planned, only an assessment of triple therapy on LDL-C change in patients with primary hypercholesterolaemia.
  Interventions: Drug: Bempedoic acid; Drug: Ezetimibe; Drug: Rosuvastatin; Drug: Atorvastatin

INTERVENTIONS:
Drug: Bempedoic acid — No drug was administered in this observational study.
Drug: Ezetimibe — No drug was administered in this observational study.
Drug: Rosuvastatin — No drug was administered in this observational study.
Drug: Atorvastatin — No drug was administered in this observational study.

SUMMARY:
Data on the real-world use and effectiveness and safety of bempedoic acid combined with both a statin and ezetimibe in clinical practice is limited. There is an increased focus on using combination therapy to lower LDL-C.

DETAILED DESCRIPTION:
The aim of the current study is to evaluate the effectiveness and safety of bempedoic acid combined with ezetimibe and either atorvastatin or rosuvastatin (hereafter defined as triple therapy) in a real-world clinical setting. No drug will be administered during this observational study.

The primary objective of the study is to evaluate the effectiveness of the triple therapy in terms of LDL-C reduction at 8 weeks.

The secondary objectives will include the following:

* Goal attainment at 8 weeks and 1 year after start of triple therapy
* Effectiveness of triple therapy in terms of LDL-C reduction at 1 year
* Effectiveness of adding bempedoic acid to statin and ezetimbe at 8 weeks and 1 year
* Effectiveness of adding bempedoic acid/ezetimibe FDC to statin in terms of LDL-C reduction at 8 weeks and 1 year
* Changes in laboratory values at 8 weeks and 1 year after start of triple therapy
* Adherence to triple therapy treatment
* Collection and recording of all adverse events occurred since initiation of triple therapy
* MACE-3 and MACE-4 (consisting of non-fatal MI, non-fatal stroke, CV-death, and coronary revascularization (for MACE-4 only)) during the year of follow-up
* Treatment changes at LMT initiation and at triple therapy initiation
* Treatment pathway from triple therapy initiation to 1-year after start of triple therapy

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent to participate
2. At least 18 years of age
3. High and very high risk patients as assessed by the physician suffering from documented primary hypercholesterolemia or mixed dyslipidemia at start of bempedoic acid treatment
4. Patients treated with:

   * bempedoic acid added to ezetimibe and rosuvastatin or atorvastatin,
   * bempedoic acid plus ezetimibe added to rosuvastatin or atorvastatin,
   * bempedoic acid plus atorvastatin or rosuvastatin added to ezetimibe
   * initiation of bempedoic acid, ezetimibe, and atorvastatin or rosuvastatin simultaneously

6) Initiation of triple therapy within a maximum of four weeks prior to inclusion 7) An untreated LDL-C value must be available within 5 years prior to the start of the triple therapy. Untreated means that the LDL-C value is not influenced by any lipid lowering therapy at the time of blood collection. Time window for not being treated as specified in the protocol.

8) No contraindications exist according to the SmPC of bempedoic acid, the respective statin and ezetimibe as per physicians' assessment 9) No concurrent participation in an interventional study (simultaneous participation in other non-interventional studies is possible) 10) Life expectancy > 1 -year

Key Exclusion Criteria:

1. Patients who have received PCSK9i monoclonal antibody treatment in the last 3 months before the start of the triple therapy exposure
2. Patients who have ever received PCSK9i-siRNA treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective data from routine clinical practice will be collected over the course of 1 year involving approximately 2000 patients across approximately 200 sites in Europe (Germany, Italy, Spain, Austria, and Belgium) treated by both specialized and non-specialized physicians in hospital and office-based settings.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Relative LDL-C change between untreated and 8 week after triple therapy start | Baseline to 8 weeks after initiation of triple therapy
  LDL-C will be assessed using a standard lipid panel blood test,

SECONDARY OUTCOMES:
Proportion of patients at ESC/EAS 2019 dyslipidemia guideline goal at 8 weeks and 1 year | Baseline to 1 year after initiation of triple therapy
  The 2019 EAS/ESC guidelines recommend treatment targets of at least a 50% reduction from baseline LDL-C levels and an LDL-C concentration below 1.8 mmol/L for patients at high and 1.4 mmol/l for patients at very high cardiovascular risk.
Relative LDL-C change between untreated and 1 year after triple therapy start | From any prior LMT exposure to 1 year after initiation of triple therapy
  LDL-C will be assessed using a standard lipid panel blood test,
Relative LDL-C change between pre-bempedoic acid/pre-FDC initiation and 8 weeks after triple therapy start | From pre-bempedoic acid/pre-FDC initiation to 8 weeks after initiation of triple therapy
  LDL-C will be assessed using a standard lipid panel blood test,
Relative LDL-C change between pre-bempedoic acid/pre-FDC initiation and 1 year after triple therapy start | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of triple therapy
  LDL-C will be assessed using a standard lipid panel blood test,
Relative change in laboratory values between triple therapy start and 8 weeks and 1 year thereafter | Baseline to 1 year after initiation of triple therapy
  Labs will be assessed using a standard panel blood test,
Patient and physician reported adherence at 8 weeks and 1 year after triple therapy start | Baseline to 1 year after initiation of triple therapy
  Adherence will be judged by the physician/patient.
Incidence of adverse events under triple therapy exposure | Baseline to 1 year after initiation of triple therapy
  Adverse events are defined as any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Proportion of patients with MACE-3 and MACE-4 events | Baseline to 1 year after initiation of triple therapy
  MACE-3 and MACE-4 events will consist of non-fatal MI, non-fatal stroke, CV-death, and coronary revascularization (for MACE-4 only).

CONTACTS AND LOCATIONS:
Locations (152):
- Austria (24):
  - Innere Medizin, Braunau am Inn
  - Innere Medizin 1, Feldkirch
  - Uniklinik Graz, Endokrinologie und Diabetes, Graz
  - Uniklinik Graz, Kardiologie, Graz
  - Innere Medizin 3 - Kardiologie, Innsbruck
  - Klinikum Wels-Grieskirchen GmbH+B18, Kepler Universitätsklinikum Gmb+
  - Innere Medizin, Klagenfurt
  - Innere Medizin, Linz
  - Kepler Universitätsklinikum GmbH Klinik für Innere Medizin 1 - Kardiologie und Internistische Intensivmedizin, Linz
  - Kardiologie-Urfahr Dr. Hönig & Dr. Gammer & Dr. Buchmayr, Linz
  - Ordination, Mattersburg
  - Landesklinikum Mistelbach - Gänserndorf, Mistelbach
  - Ordination Dr. med. univ. Evelyn Fließer-Görzer, Saint Stefan Bei Graz
  - Praxis Gesundheitszentrum Moos 15 (Praxis Prof. Lichtenauer), Salzburg
  - DOZ (Dialyse- und Ordinationszentrum) Privatklinik Wehrle-Diakonissen, Salzburg
  - Klinik Landstrasse, Kardiologie, Vienna
  - Ordination Univ.-Prof. Dr. Kurt Huber, Vienna
  - Zentrum für Klinische Studien Dr. Hanusch GmbH, Vienna
  - AKH Wien, Vienna
  - Meduni Wien, Endokrinologie und Diabetes, Vienna
  - Meduni Wien, Kardiologie, Vienna
  - Clinic Hietzing, Vienna
  - Herzzentrum 18, Vienna
  - Karl Landsteiner Institut für kardiovaskuläre und intensivmedizinische Forschung c/o Abteilung für Kardiologie, Klinik Floridsdorf, Vienna
- Belgium (14):
  - Azorg, Aalst
  - UZA (Antwerp University Hospital), Antwerp
  - A.Z. KLINA Brasschaat, Brasschaat
  - Algemeen Ziekenhuis Sint-Jan Oostende, Bruges
  - Z.O.L - Campus St. Jan, Genk
  - Az Sint Lucas, Ghent
  - CHR Huy, Huy
  - AZ Groeninge Kortrijk, Kortrijk
  - Pôle hospitalier Jolimont, La Louvrière
  - JAN YPERMAN Ziekenhuis, Leper
  - CHR Citadelle de Liège, Liège
  - AZ Delta, Roeselare
  - AZ Glorieux, Ronse
  - CHU UCL Mont-Godinne, Yvoir
- Germany (37):
  - Praxis für Kardiologie Aachen, Aachen
  - Klinikum Ahaus, Ahaus
  - Praxis W. Almohamed, Alsfed
  - Zentrum für klinische Studien Bad Homburg, Bad Homburg
  - Dialysezentrum Hellersdorf Mitte, Berlin
  - Lipidambulanz Charite Campus Virchow, Berlin
  - MEDICLIN Reha-Zentrum Spreewald, Burg
  - Kardiologische Gemeinschaftspraxis Flemmingstr., Chemnitz
  - Klinik Detmold, Detmold
  - Praxis Dr. Methfessel, Dresden
  - Cardiologicum Dresden, Dresden
  - Herz- und Gefäßmedizin Goslar, Goslar
  - ndgl.; viele Kombinationstherapien, Gräfenhainichen
  - Praxis, Greiz
  - Kardiologie am Tibarg, Hamburg
  - HPK Heidelberger Praxisklinik, Heidelberg
  - Uni-Klinik Heidelberg, Heidelberg
  - Kardiopraxis, Kaiserslautern
  - GK Mittelrhein, Koblenz
  - Klinikum Konstanz, Konstanz
  - Universitätsklinikum Leipzig, Leipzig
  - DRK Krankenhaus Lichtenstein Gemeinnützige GmbH, Lichtenstein
  - Cardio Centrum Ludwigsburg, Ludwigsburg
  - Kardiopraxis, Mainz
  - Kardiologische Praxis Markkleeberg, Markkleeberg
  - Kardiologie Gem. Praxis Dres Reiff/Linse/Haj-Yehia/Specking, Moers
  - Praxis Dr. Norbert Schön, Mühldorf A. Inn
  - Kardiologische Gemeinschaftpraxis Papenburg, Papenburg
  - Kardiologische Gemeinschaftspraxis Papenburg, Papenburg
  - Hausärztlich-kardiologisches MVZ,,Am Felsenkeller" GmbH, Pirna
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam
  - Lipidambulanz Uniklinikum Regensburg, Regensburg
  - Parkkardiologie, kard. Gemeinschaftspraxis, Stanhsdorf B. Berlin
  - BBT Trier, Trier
  - Diabetologische Schwerpunktpraxis, Trier
  - Herzklinik, Ulm
  - Dialysezentrum Hofaue, Wuppertal
- Italy (41):
  - Ente Ecclesiastico "Miulli", Acquaviva delle Fonti
  - INRCA, Ancona
  - AO Moscati, Avellino
  - Osp. "San Paolo", Bari
  - Ospedale di Bolzano, Bolzano
  - Spedali Civili di Brescia, Brescia
  - Osp. santo spirito, Casale Monferrato
  - Ospedale Sant'Anna e san Sebastiano, Caserta
  - Osp. SS Annunziata, Chieti
  - PO Nuovo Umberti I, Enna
  - Osp. Sant'Anna di Cona, Ferrara
  - Policlinico "Riuniti", Foggia
  - Policlinico San Martino, Genova
  - Osp della Misericordia, Grosseto
  - Osp. "Vito Fazzi", Lecce
  - Ospedale Mater Salutis, Legnagno
  - Spedali Riuniti, Livorno
  - Ospedale di Mantova, Mantova
  - Policlinico G. Martino, Messina
  - IRCCS Monzino, Milan
  - IRCCS Galeazzi Sant'Ambrogio, Milan
  - Policlinico Modena, Modena
  - AO Cardarelli, Napoli
  - Policlinico Federico II, Napoli
  - AOU Vanvitelli, I Policlinico, Napoli
  - Policlinico P. Giaccone, Palermo
  - ICS Maugeri, Pavi
  - S. Maria della Misericordia, Perugia
  - Ospedale PederzoliItlit, Peschiera
  - Cisanello, Pisa
  - Osp. Santa Maria delle Croci, Ravenna
  - Osp infermi di rivoli, Rivoli
  - Policlinico Tor Vergata, Roma
  - Ospedale Pertini, Roma
  - Ospedale Sant'Andrea, Roma
  - Policlinico Umberto I, Rome
  - Molinette Università to, Torino
  - Ospedale Mauriziano, Torino
  - Osp. di Cattinara, Trieste
  - Ospedale di Portogruaro, Venezia
  - AOUI Verona, Verona
- Spain (36):
  - H. Univers. De Albacete, Albacete
  - Hospital General Universitario Dr. Balmis, Alicante
  - H. General de Elche, Alicante
  - Hospital Universitario de San Juan, Alicante
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitario de Burgos, Burgos
  - H. Univ. Puerta del Mar, Cadiz
  - H. Punta de Europa, Cadiz
  - Hospital Universitario Puerto Real, Cadiz
  - Sierrallana Hospital, Cantabria
  - H. Univ. Reina Sofía, Córdoba
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - H. Univ. De Cabueñes, Gijón
  - H. Virgen de las Nieves, Granada
  - H. Juan Ramón Jiménez, Huelva
  - Hospital Universitario Médico-Quirúrgico de Jaén, Jaén
  - Hospital Universitario de Gran Canarias Dr. Negrín, Las Palmas de GC
  - Hospital de León, León
  - Hospital San Pedro, Logroño
  - H. Costa del Sol, Marbella (Málaga)
  - H. Virgen de la Victoria, Málaga
  - Hospital Serranía de Ronda, Málaga
  - Hospital General Universitario Reina Sofía, Murcia
  - H. Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Son LLatzer, Palma de Mallorca
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital de Segovia, Segovia
  - Hospital General Universitario de Toledo, Toledo
  - H. Clínico Univ. De Valencia, Valencia
  - Consorcio Hospital General Univ de Valencia, Valencia
  - Hospital La Fe, Valencia
  - Hospital Universitario de Álava, Vitoria-Gasteiz
  - Hospital Clinico Universitaro Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No